Official title: EVALUATION OF A RESPIRATORY MUSCLE TRAINING PROGRAM RESTRICTING NASAL BREATHING WITH FEELBREATHE® DEVICE IN COPD PATIENTS

Date of the document: 04-04<sup>th</sup>-2017

# Background

The benefits of pulmonary rehabilitation programs (RP) in chronic obstructive pulmonary disease (COPD) patients have been shown and are recognized as an effective tool for improving dyspnea, exercise tolerance and quality of life in all the guidelines(1)(2)(3).

Inspiratory muscles training (IMT) has been used as a complement added to the supervised pulmonary RP and some studies have shown an improvement in the inspiratory muscles strength, tolerance to exercise (Oxygen uptake efficiency slope), dyspnea and distance walked in the six minutes walking test (6MWT) after a inspiratory muscles training program in patients with COPD (4).

The Feelbreathe® device, tested in our study can be used in static and dynamic situations (5) and is a nasal ventilatory flow restriction device made by a strip of hypoallergenic material (3M Spain, S.A. Medical Specialties / O.E.M.) that is placed and adhered under the nostrils impairing the free pass of air through the nose by producing resistance to flow. The Feelbreathe® device (FB) has been authorized by the Spanish Agency for Medicines and Health Products for application on COPD patients (Expedient 521/15/EC. AEMPS-Madrid-Spain-Patent N°: P200902402).

Previous studies have shown that an increased airflow resistance while breathing nasally, during exercise, increases the breathing effort (6) which may potentially improve the exercise tolerance (7) and energy efficiency (8). In healthy subjects FB has shown changes in lung ventilation, gas exchange and heart rate during exercise with improvements on ventilatory efficiency (9).

So, the objective of this study was to assess the effects of a nasal restriction device for inspiratory muscle training adding to a rehabilitation program on exercise capacity (Oxygen uptake efficiency slope), quality of life, dyspnea and inspiratory muscle strength in stable COPD patients.

#### STUDY PROTOCOL AND STATISTICAL ANALYSIS PLAN

## **Participants**

Subjects were recruited from the Pneumology outpatient of the University Hospital Puerta del Mar in Cádiz (Spain). Consecutive patients were screened by reviewing their charts and by interview. Inclusion criteria were diagnosis of COPD according to guidelines criteria (1) (10) with moderate or severe airflow obstruction (GOLD 2 or 3)(10), dyspnea grade 2 or greater by mMRC scale and a stable clinical condition for at least 2 months. Exclusion criteria were poor compliance, treatment with oxygen therapy or non-invasive mechanical ventilation, CO<sub>2</sub> retention, medical conditions that can produce or increase dyspnea on exercise in addition to COPD (cardiovascular, metabolic or other respiratory diseases) or osteoarticular or neuromuscular diseases that may limit the correct performance of the 6MWT. A total of 36 patients were included in this study.

Written informed consent was obtained from all patients before starting the study. This clinical trial received ethical approval from the Ethics Committee University Hospital Puerta del Mar and met the requirements of the Declaration of Helsinki.

# Design

Participants were randomly assigned according to a computer-generated randomization table to three groups: 1) those who participated in the supervised RP using the Feelbreathe® device (FB group), 2) those who participated in the supervised RP with oronasal breathing without Feelbreathe® device (ONB group) and, 3) those included in the control group (CG) which received standard medical recommendation for patients with COPD.

Demographic and clinical data were recorded. Dyspnea was assessed by the modified Medical Research Council (mMRC) dyspnea questionnaire (11) and quality of life by the COPD Assessment Test (CAT) questionnaire (12). Spirometry was performed according to American Thoracic Society criteria (13)(14) {Formatting Citation (Spirometer CPX, Cardinal Health, Hoechberg, Germany). Then, they performed a resting electrocardiogram (QRS Universal ECG, QRS, Plymouth, MN, USA). P<sub>Imax</sub> was measured during a maximal, static inspiratory effort measured at the mouth (Micro RPM, Micro Medical Ltd., Chatham, Kent, UK). P<sub>Imax</sub> was recorded as the highest value averaged over 1s from three maneuvers that varied by less than 10% and was measured based on three maximal reproducible respiratory efforts. Then, an incremental test on treadmill (Technogym Run Race 1400HC, Gambettola, Italy) was performed to determine the VO<sub>2</sub>peak (Circuit Spirometry Vmax 29C, Sensormedics, USA). While performing the tests, the cardiac response was measured every 10s (JECG 12 Canal, Friedberg, Alemania). Blood oxygen saturation percentage (Ear oximeter, Hewlett-Packard 47201A, Corvallis, EEUU) and respiratory gas exchange were measured every 5 sand breath by breath respectively, throughout the test. Finally, one week apart, the patients performed the 6MWT according to the ATS guideline (15).

All tests were performed according to a standardized protocol before starting the training and 2 days after its completion.

#### Training program

Participants carried out a supervised RP for 8 weeks, 3 days per week. The training sessions lasted 60 minutes and included a warning up phase, a main phase and a recovery phase. After each session, Borg's perceived exertion was measured. The RP included aerobic exercise on cycle ergometer and on treadmill (progressing since 10' to 30' and since 40 to 75% of the reserve heart rate (RHR) or 6-7 score based on Borg's perceived exertion), strengthening of lower and upper limb muscles groups, breathing exercises (pursed lip breathing, diaphragmatic and abdominal breathing and diaphragmatic mobility) and finally stretching exercises.

In the FB group, for restricted nasal breathing, at the beginning of the training program, the small size device was used (4 mm). The size of the device was progressively increasing according to the patient adaptation to the 5 or 6 mm device,

depending on the score on Borg's perceived exertion scale. If the patient has a score under 4 after the RP sessions the size of the FB device was increased.

FB was placed under the nostrils, using sterile gloves and assessing the patient did not have mucus or injuries. The device was used during the RP and patients were invited to have a physiological breathing by nasal inspirations and mouth expirations.

### **Statistical Analysis**

Descriptive data of the participants are expressed as mean  $\pm$  standard deviation or number and percentage for continuous and categorical variables respectively. Percentage of change ( $\%_{Change}$ ) for each variable was calculated as:

%<sub>Change</sub> = (mean(Post-test value) – mean(Pre-test value) / mean(Pre-test value)) \* 100

Differences among RP (between differences) and between pre- and post RP tests within each breathing condition (within differences) were analysed using a Bayesian hierarchical model. 6MWT distance, P<sub>Imax</sub> and CAT were considered as continuous variables while mMRC dyspnea was treated as an ordinal variable. To analyse differences at baseline only a categorical variable indicating the RP (GC, ONB or FB) was introduced in the model as predictor. However, to analyse both between and within differences RP, time (pre- or post-PR) and their interaction were introduced as predictor variables. Due to the sample size in our study we choose to analyse our data using Bayesian inference since it has proven to be a proper method of statistical inference for small sample size (16)(17). Inference was performed based on the 95% credible interval (95% CrI) which contains a range of values where we can be 95% certain that the true value lie given the data at hand and the model fitted. The Bayesian hierarchical model was fitted using the package brms for the R programming language for statistical computing and graphics (18). All parameters estimated showed a good convergence with values of  $\hat{R} = 1$  and number of effective sample size > 1000. Further analysis can be found in the supplemental file while the code and the dataset to replicate it are stored in https://github.com/JorgeDelro/COPD 2 1.

### References

- 1. Miravitlles M, Soler-Cataluña JJ, Calle M, Molina J, Almagro P, Quintano JA, et al. Guía española de la enfermedad pulmonar obstructiva crónica (GesEPOC) 2017. Tratamiento farmacológico en fase estable. Arch Bronconeumol. 2017 Jun;53(6):324–35.
- 2. GlobalStrategy for the diagnosis, management, and prevention of Chronic Obstructive Pulmonary Disease (2019 Report) [Internet]. 2019. Available from: www.goldcopd.org
- 3. Celli BR, MacNee W, Agusti A, Anzueto A, Berg B, Buist AS, et al. Standards for the diagnosis and treatment of patients with COPD: a summary of the ATS/ERS position paper. Eur Respir J. 2004;23(6):932–46.
- 4. Lötters F, van Tol B, Kwakkel G, Gosselink R. Effects of controlled inspiratory muscle training in patients with COPD: A meta-analysis. Eur Respir J. 2002;20(3):570–6.
- 5. González Montesinos JL, Costa Sepúlveda JL, Fernández Santos J, Gómez Espinosa de los Monteros R, Mora Vicente J, Castro Piñero J y, et al. Dispositivo de Restricción y Filtrado del Flujo Ventilatorio Nasal. P200902402, 2011. p. 1–4.

- 6. Morton AR, King K, Papalia S, Goodman C, Turley KR, Wilmore JH. Comparison of maximal oxygen consumption with oral and nasal breathing. Aust J Sci Med Sport. 1995;27:51–5.
- 7. Bailey SJ, Romer LM, Kelly J, Wilkerson DP, DiMenna FJ, Jones AM. Inspiratory muscle training enhances pulmonary O(2) uptake kinetics and high-intensity exercise tolerance in humans. J Appl Physiol. 2010;109:457–68.
- 8. Illi SK, Held U, Frank I, Spengler CM. Effect of respiratory muscle training on exercise performance in healthy individuals: A systematic review and meta-analysis. Vol. 42, Sports Medicine. 2012. p. 707–24.
- 9. González-Montesinos JL, Ponce-González JG, Vicente-Campos D, López-Chicharro J, Fernández-Santos JR, Vaz-Pardal C, et al. Efectos de un dispositivo de restricción ventilatoria nasal sobre la ventilación pulmonar e intercambio gaseoso durante el ejercicio en personas sanas. Nutr Hosp. 2016;33(2):444–50.
- 10. Vogelmeier CF, Criner GJ, Martinez FJ, Anzueto A, Barnes PJ, Bourbeau J, et al. Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease 2017 Report. GOLD Executive Summary. Am J Respir Crit Care Med [Internet]. 2017 Mar 1 [cited 2019 Apr 5];195(5):557–82. Available from: http://www.ncbi.nlm.nih.gov/pubmed/28128970
- 11. Cotes JE, Chinn DJ. MRC questionnaire (MRCQ) on respiratory symptoms. Vol. 57, Occupational Medicine. 2007. p. 388.
- 12. Jones PW, Harding G, Berry P, Wiklund I, Chen W-H, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648–54.
- 13. Culver BH, Graham BL, Coates AL, Wanger J, Berry CE, Clarke PK, et al. Recommendations for a Standardized Pulmonary Function Report. An Official American Thoracic Society Technical Statement. Am J Respir Crit Care Med. 2017 Dec;196(11):1463–72.
- 14. Redlich CA, Tarlo SM, Hankinson JL, Townsend MC, Eschenbacher WL, Von Essen SG, et al. Official American Thoracic Society technical standards: spirometry in the occupational setting. Am J Respir Crit Care Med. 2014;189(8):983–93.
- 15. ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul;166(1):111–7.
- 16. van de Schoot R, Broere JJ, Perryck KH, Zondervan-Zwijnenburg M, van Loey NE. Analyzing small data sets using Bayesian estimation: the case of posttraumatic stress symptoms following mechanical ventilation in burn survivors. Eur J Psychotraumatol. 2015 Dec;6(1):25216.
- 17. van de Schoot R, Sijbrandij M, Depaoli S, Winter SD, Olff M, van Loey NE. Bayesian PTSD-Trajectory Analysis with Informed Priors Based on a Systematic Literature Search and Expert Elicitation. Multivariate Behav Res. 2018 Mar;53(2):267–91.
- 18. Bürkner P-C. brms: An R Package for Bayesian Multilevel Models Using Stan. J Stat Softw. 2017;80(1).